CLINICAL TRIAL: NCT01388751
Title: Night Splinting After 6 to 8 Weeks of Continuous Splinting for Mallet Finger
Brief Title: Mallet Finger Splinting Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David C. Ring, MD, Principal Investigator; Director of Research, Hand Service, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008P001506
Record Dates: First submitted 2011-07-05; First posted 2011-07-07 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Mallet Finger
Keywords: Mallet Finger splinting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- no night splinting (No Intervention)
- night splinting (Active Comparator): Night Splinting for 4 weeks after removal of initial cast
  Interventions: Procedure: night splinting

INTERVENTIONS:
Procedure: night splinting — splint finger at night for 4 weeks
  Arms: night splinting

SUMMARY:
Do patients that night splint for 1 month after 6-8 weeks of continuous splinting for a mallet injury have the same extensor lag 4 months after initiating treatment as patients that do not perform night splinting?

Secondary Question: Is night splinting a predictor of DASH score or patient satisfaction (on a 5-Point Likert scale)?

ELIGIBILITY:
Inclusion Criteria:

* All adult, English-speaking patients in the practice of Dr. Jesse Jupiter, Dr. Chaitanya Mudgal, or Dr. David Ring electing splint treatment for mallet deformity will be invited to enroll on their follow-up visit 6-8 weeks after initiating splint treatment.

Exclusion Criteria:

1. Open lesions
2. Mallet fracture more than 2 weeks old
3. Mallet fracture with subluxation of the distal interphalangeal joint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-11; Primary Completion 2012-05 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Extensor Lag | 4 months
  Null Hypothesis:
  Patients that night splint for 1 month after 6-8 weeks of continuous splinting for a mallet injury have the same extensor lag 4 months after initiating treatment as patients that do not perform night splinting.

SECONDARY OUTCOMES:
DASH score | 4 months
  Secondary Study Questions:
  Is night splinting a predictor of DASH score or patient satisfaction (on a 5-Point Likert scale)?

CONTACTS AND LOCATIONS:
Overall Officials: David Ring, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States